CLINICAL TRIAL: NCT00035997
Title: An Open-label Trial on the Effect of I.V. Zoledronic Acid 4 mg on Bone Mineral Density in Hormone Sensitive Prostate Cancer Patients With Bone Metastasis
Brief Title: Open-label Trial on the Effect of I.V. Zoledronic Acid 4 mg on Bone Density in Hormone Sensitive Prostate Cancer Patients With Bone Metastasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EUS24; US24
Record Dates: First submitted 2002-05-07; First posted 2002-05-08 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Prostate Cancer
Keywords: Hormone-sensitive Prostate Cancer; Prostate Cancer; Bone Metastasis
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zometa

SUMMARY:
The purpose of this trial with Zometa is to investigate the effect ZOMETA 4 mg (zoledronic acid for injection in 100mg solution ) has in preventing associated bone loss in prostate cancer patients with bone metastasis when administered in conjunction with hormonal cancer therapy. This trial will seek to determine the effect of ZOMETA in stabilizing and increasing bone mineral density in these patients.

This prospective, open-label, single arm, multicenter study will enroll approximately 200 prostate cancer patients with a history of at least one documented bone lesion documented by bone scan or radiograph. Patients must already be receiving hormone therapy and meet the following additional criteria:

* 18 years of age or older
* Histologically confirmed diagnoses of prostate cancer
* Confirmed objective evidence of metastatic bone disease as evidenced by bone scan or radiograph
* Received or will receive hormonal treatment also know as androgen deprivation therapy with an LHRH agonist or other hormonal treatments

Throughout the course of this 12-month trial, patients will be identified based on the duration of established hormonal treatment at the time of enrollment. Each patients duration of participation will be up to 56 weeks including a 4 week screening, 48 week treatment and a 4 week follow up.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent
* Age > 18 years
* Histologically confirmed diagnosis of carcinoma of the prostate
* Objective evidence of metastatic disease to the bone as evidenced by bone scan or radiograph at any point since their diagnosis of prostate cancer
* Currently receiving, or will begin receiving, hormonal therapy with an LHRH agonist or other hormonal treatments for either < 6 months or > 6 months
* ECOG performance status of 0, 1, or 2

Exclusion criteria:

* Patients who are hormone sensitive without metastatic disease to the bone
* Patients who are hormone refractory typically defined as two or three consecutive increases in PSA measured at least one month apart while on hormone therapy
* Patients who are not treated with LHRH agonist or other hormonal treatments
* Patients who are currently receiving diethylstilbestrol (DES) or PC-SPES
* Patients with another nonmalignant disease which would confound the evaluation of primary endpoints or prevent the patient complying with the protocol.
* Patients with abnormal renal function as evidenced by either a serum creatinine greater than 2 mg/dL or by a calculated creatinine clearance of 60 ml/minute or less
* Corrected (adjusted for serum albumin) serum calcium concentration < 8.0 mg/dl (2.00 mmol/L)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2002-04; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Changes in bone mineral density of the lumbar spine (L2-L4) at 12 months

SECONDARY OUTCOMES:
Changes in biochemical markers of bone turnover over 12 months
Changes in bone mineral density of the total hip at 12 months
Time to first skeletal-related event
Overall safety measured by adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Scott L. Pescatore, PharmD., Study Director — Novartis
Locations (56):
- United States (56):
  - Norwood Clinic, Birmingham, Alabama
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Advanced Urology Medical Center, Anaheim, California
  - Urology Associates of Central CA, Fresno, California
  - Center for Urological Research, La Mesa, California
  - Atlantic Urological Medical Group, Long Beach, California
  - Advanced Urology Medical Offices, Los Angeles, California
  - Advanced Urology Medical Office, Los Angeles, California
  - Boulder Medical Center, Boulder, Colorado
  - Urology Associates, P.C., Denver, Colorado
  - Atlantic Urological Associates, Daytona Beach, Florida
  - Southwest Florida Urologic Association, Fort Myers, Florida
  - Diagnostic Clinic, Largo, Florida
  - DMI Health Care Group, Inc., Largo, Florida
  - Marvin Stein, MD, Margate, Florida
  - Miami Cancer Institute, Miami, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Florida Foundation for Healthcare Research, Ocala, Florida
  - Urology Associates of Northeast Florida, PA, Orange Park, Florida
  - Winter Park Urology Associates, Orlando, Florida
  - Pinellas Urology, Inc., St. Petersburg, Florida
  - Southeastern Urological Center, Tallahassee, Florida
  - Georgia Urology Research Institute, Atlanta, Georgia
  - Ball Memorial Hospital, Muncie, Indiana
  - Urological Associates PC, Davenport, Iowa
  - Drs. Werner, Murdock and Francis PA Urology Associates, Greenbelt, Maryland
  - Urology Associates of Middlesex County, Inc., Marlborough, Massachusetts
  - Lakeside Urology, P.C., Saint Joseph, Michigan
  - Millennium Medical Center, Southfield, Michigan
  - Kansas City Urology Care, Kansas City, Missouri
  - The Prostate Center of Greater St. Louis, St Louis, Missouri
  - American Academy of Urology, Las Vegas, Nevada
  - Urological Surgical Associates, Edison, New Jersey
  - UroResearch, LLC, Morristown, New Jersey
  - Shaukat M. Qureshi, MD, Pennsville, New Jersey
  - Urology Associates, Stratford, New Jersey
  - Associates in Urology, LLC, West Orange, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - Urological Surgeons of Long Island PC, Garden City, New York
  - Kingston Urological Assoc., Kingston, New York
  - Cary Urology, P.A., Cary, North Carolina
  - Matrix Research, LLC, Greenville, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Southwest Urology, Parma, Ohio
  - Roger N. Andrews, MD Inc., Arcadia, Pennsylvania
  - Urologic Surgery, PC, Bala-Cynwyd, Pennsylvania
  - James W. Thompson, MD Ltd., Bryn Mawr, Pennsylvania
  - Urology Institute of Pittsburgh, Monroeville, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Center for Urologic Care of Berks County, West Reading, Pennsylvania
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Urology Center of the South P.C., Germantown, Tennessee
  - Murfreesboro Medical Clinic, Murfreesboro, Tennessee
  - Urology Associates, PA, Nashville, Tennessee
  - Research Across America, Carrollton, Texas
  - CAMC Clinical Trials, Charleston, West Virginia